CLINICAL TRIAL: NCT05443217
Title: Intestinal and Oral Microbiota Signatures of Clinical Response and Adverse Events in HCC Treated With Systemic Therapies
Brief Title: Relationship Between Microbiota and Prognosis of Hepatocellular Carcinoma(HCC) After Systemic Treatments
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Qilu Hospital of Shandong University (Other); Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Gang Chen, MD, Clinical Professor, Principal Investigator, First Affiliated Hospital of Wenzhou Medical University
Other Study IDs: microbiota
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Liver Cancer; Microbiota; Adverse Event; Prognosis; Efficacy
Keywords: HCC; microbiota; Adverse Event; prognosis; efficacy
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fecal sample, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with response to systemic therapies
  Interventions: Diagnostic Test: questionnaire survey
- patients with no response to systemic therapies
  Interventions: Diagnostic Test: questionnaire survey

INTERVENTIONS:
Diagnostic Test: questionnaire survey — All patients received lifestyle questionnaire, physical performance, and imaging evaluation before treatment.

SUMMARY:
By tracking the short-term and long-term results of HCC patients treated with systemic therapies,the difference of microbiota between responded patients and non-responded patients was analyzed, and the correlation between gut and oral microbiota and short-term and long-term results was explored, so as to improve people's awareness of microbiota and pay attention to its prevention and treatment.

DETAILED DESCRIPTION:
The investigators consecutively admit patients the questionnaire and collect the fecal. And by tracking the short-term and long-term outcomes of HCC patients treated with systemic therapies,the difference of gut microbiota between responded patients and non-responded patients is analyzed, and the correlation between gut and oral microbiota and short-term and long-term results is explored.Adverse events (AE) are recorded using the National Cancer Institute's Common Terminology Criteria for Adverse Events (version 4.0).Tumor response is mainly evaluated by experienced hepatologists using radiological method within 4-12 weeks after treatments according to the RECIST 1.1 and Modified Response Evaluation Criteria in Solid Tumors (mRECIST).Overall survival (OS) and Progression-free survival (PFS) are recorded.

ELIGIBILITY:
Inclusion Criteria:

* clinically or pathologically diagnosed HCC
* didn't receive prior anti-tumor treatments
* didn't receive prior antibiotics
* Eastern Cooperative Oncology Group performance status (ECOG-PS) 0-1
* Child-Pugh score of ≤7
* complete clinical and follow-up information.

Exclusion Criteria:

* combined with other malignancies
* receive surgical treatment
* lost follow-up
* Child-Pugh score of>7
* uncompleted clinical and follow-up information
* overall survival less than 1 month
* receive prior antibiotics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with unresectable HCC who received systemic therapies
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Post-treatment adverse events | 3 months
  Post-treatment complications are recorded
Long-term outcomes after treatment | 1 year
  Overall survival and progression-free survival

SECONDARY OUTCOMES:
Objective response rate | 3 months
  Tumor response

CONTACTS AND LOCATIONS:
Locations (1):
- Gang Chen, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCulloch JA, Davar D, Rodrigues RR, Badger JH, Fang JR, Cole AM, Balaji AK, Vetizou M, Prescott SM, Fernandes MR, Costa RGF, Yuan W, Salcedo R, Bahadiroglu E, Roy S, DeBlasio RN, Morrison RM, Chauvin JM, Ding Q, Zidi B, Lowin A, Chakka S, Gao W, Pagliano O, Ernst SJ, Rose A, Newman NK, Morgun A, Zarour HM, Trinchieri G, Dzutsev AK. Intestinal microbiota signatures of clinical response and immune-related adverse events in melanoma patients treated with anti-PD-1. Nat Med. 2022 Mar;28(3):545-556. doi: 10.1038/s41591-022-01698-2. Epub 2022 Feb 28. PMID 35228752
- [Background] Zheng Y, Wang T, Tu X, Huang Y, Zhang H, Tan D, Jiang W, Cai S, Zhao P, Song R, Li P, Qin N, Fang W. Gut microbiome affects the response to anti-PD-1 immunotherapy in patients with hepatocellular carcinoma. J Immunother Cancer. 2019 Jul 23;7(1):193. doi: 10.1186/s40425-019-0650-9. PMID 31337439